CLINICAL TRIAL: NCT00113217
Title: A Phase II Neoadjuvant Clinical Trial to Evaluate the Efficacy of Recombinant Humanized Monoclonal Anti-VEGF Antibody rhuMab VEGF (Bevacizumab) for Renal Cell Carcinoma
Brief Title: Neoadjuvant Clinical Trial to Evaluate the Efficacy of Bevacizumab for Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0982
Record Dates: First submitted 2005-06-06; First posted 2005-06-07 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer
Keywords: Renal Cell Carcinoma; Kidney Cancer; Bevacizumab; Avastin; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab (Experimental): 10 mg/kg intravenous (IV) Day 1 of 14-day cycle.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg IV on day 1 of each 14-day cycle.
  Other Names: Avastin

SUMMARY:
The goal of this clinical research study is to learn if bevacizumab (Avastin®) can control metastatic renal cell carcinoma (RCC). The safety of the treatment will also be studied.

Objectives:

Primary:

1. To assess the efficacy of neoadjuvant therapy of bevacizumab by evaluating time to progression.
2. Toxicities of therapy with bevacizumab in RCC.

Secondary:

Clinical:

1. Response rate
2. Duration of response
3. Overall Survival

Preclinical:

1. Serum and plasma levels of matrix metalloproteinase 9 (MMP-9) and MMP-2, Interleukin 6 (IL-6), vascular endothelial growth factor (VEGF), and Basic Fibroblast Growth Factor (bFGF) pre- and post- therapy (optional studies).
2. Tissue expression of Phospho-epidermal growth factor receptor (EGFR), VEGF, vessel count CD31/34, AKT and Phospho-AKT, mitogen-activated protein kinase (MAPK), transforming growth factor-alpha (TGF-alpha), phospho-STAT3 and TUNEL post therapy (optional studies).
3. complementary DNA (cDNA) microarray analysis of tissue post-therapy (optional studies).
4. Tissue expression of tumor infiltrating lymphocytes and tumor antigens
5. Pathological response rate in primary tumor.
6. To evaluate the Single Nucleotide Polymorphisms (SNP) patterns in nephrectomy specimens from patients participating in the study.

DETAILED DESCRIPTION:
Bevacizumab is a drug that binds to and inhibits VEGF, a blood-vessel stimulating agent with unusually high levels in kidney cancer. This drug may decrease the growth of kidney cancer.

Every two week study cycle, you will receive a dose of bevacizumab intravenously (through a needle in your vein). The first bevacizumab dose will be given over 90 minutes as a continuous IV infusion. If the first dose is tolerated without any side effects related to the intravenous (IV) infusion, the second dose may be delivered over 60 minutes. If the 60 minute infusion is tolerated, all doses of bevacizumab after that may be given over 30 minutes. If you experience infusion-related side effects with the 60 minute infusion, all doses after that will be given over 90 minutes. If you experience infusion-related side effects with the 30 minute infusion, all doses after that will be given over 60 minutes. Other drugs, including Tylenol and Benadryl, may be given before, during, and after the therapy to help prevent or ease side effects. These drugs may be given either by mouth or through an IV line.

During treatment, blood samples (about 1 1/2 tablespoons) will be taken once per 2 week cycle. Urine samples will be taken at the beginning of each cycle. At around 56 days into treatment, tumors will be measured using X-rays or other scans.

Treatment will be stopped after 56 days of therapy. In this first phase, you will receive 4 doses of bevacizumab.

If the cancer is stable or shrinks while on bevacizumab for the first 56 days, and you tolerated the treatment well, you will undergo surgery to remove your kidney tumor. Surgery will be scheduled at least 4 weeks after your last dose of bevacizumab. Approximately 4 weeks after surgery, you will undergo repeat CT scans. If your cancer is stable or continuing to shrink, you will restart treatment with bevacizumab. You will continue to have tumor measurements by scans around every 56 days (8 weeks) while receiving bevacizumab, if your initial scans showed evidence of tumor presence. However, If your tumor grew substantially during the operative period, i.e. between the first set of scans on or around day 56 and the scans performed after surgery, you will be taken off the study, and other treatments will be offered to you.

If the cancer grew while on bevacizumab for the first 56 days, you will undergo surgery to remove your kidney tumor. Surgery will be scheduled at least 4 weeks after your last dose of Bevacizumab. After surgery, you will not continue on bevacizumab. Once you recover from surgery, your doctor may recommend a different drug therapy to treat your cancer.

In some circumstances, after the first 56 days of therapy with bevacizumab, your doctors may decide that it is not possible or helpful for your kidney to be removed because of progression of your cancer rendering such an operation either not feasible or inappropriate for your care. In that case, your doctors may recommend a different drug therapy for your cancer, and you will not continue on bevacizumab.

You may be taken off study if your disease progresses or intolerable side effects occur.

If you are taken off study, you will have repeat scans, a physical examination, blood testing (about 2 tablespoons), urine testing, and an ECG. If you have elevated blood pressure or excess protein in your urine, you will be asked to come back every 2 months for repeat blood pressure testing and urine testing until these levels fall to a normal range, for up to one year.

This is an investigational study. Avastin is commercially available and approved by the FDA for metastatic colorectal cancer and small cell lung cancer. The drug is experimental and authorized for research purposes only in renal cell carcinoma. Up to 50 participants will take part in this study. All will be enrolled at The University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed clear cell metastatic RCC who are eligible for cytoreductive nephrectomy.
* Patients must have measurable disease, defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures greater than or equal to 20 mm with conventional techniques or greater than or equal to 10 mm with spiral computed tomography (CT) scan. This does not include primary tumors, which will be removed.
* The Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1
* Female patients of childbearing potential (i.e. premenopausal, no hysterectomy) must have a normal plasma beta human chorionic gonadotropin (bHCG) within 24 hours prior to enrolling in the study due to the possible teratogenic effect. Patients with an elevated bHCG will undergo appropriate evaluation to rule out pregnancy (i.e. referral to Gyn service, pelvic ultrasound) and if pregnancy is ruled out and elevated bHCG is determined to be of tumor origin, patients will be permitted to proceed on study.
* Patients of child fathering or childbearing potential must agree to practice a form of medically acceptable birth control while on study, i.e. condoms.
* Patients must give written informed consent prior to initiation of therapy, in keeping with the policies of the institution. Patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy. The only approved consent is attached to this protocol.
* Patients must have ability to comply with study and/or follow-up procedures.
* Patients must have adequate organ and marrow function within 14 days as defined below: absolute neutrophil count >/=1,500/micro platelets >/= 75,000/micro Hgb > 9.0 g/dL (may be transfused or receive epoetin alfa permitted) total bilirubin </= 2.0 mg/dL albumin > 3.0 g/dL serum creatinine </= 2.0 mg/dL aspartate aminotransferase (AST or SGOT) and/or alanine aminotransferase (ALT or SGPT) </= 2.5 * upper limit of normal (ULN), no liver metastases AST(SGOT) and/or ALT (SGPT) </= 5 * ULN, liver metastases present.

Exclusion Criteria:

* Patients must not have organ allografts.
* Patients must not have had major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study (other than defined by protocol); or fine needle aspirations or core biopsies within 7 days prior to Day 0.
* No prior malignancy is allowed, except for non-melanoma skin cancer, in situ carcinoma of any site, or other cancers for which the patient has been adequately treated and disease free for 5 years.
* Patients must not have received any systemic anticancer therapy. Radiation therapy is allowed if >/= 2 weeks from study drug administration.
* Patients must not be scheduled to receive another experimental drug while on this study. Patients are permitted to be on concomitant bisphosphonates and megestrol acetate.
* Patients must not have a primary brain tumor (excluding meningiomas other benign lesions), any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, or history of stroke within the past 5 years.
* History of serious systemic disease, including myocardial infarction or unstable angina within the last 12 months, history of hypertensive crisis or hypertensive encephalopathy, uncontrolled hypertension (blood pressure of >140/90 mmHg on medication), New York Heart Association (NYHA) Grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), significant vascular disease or symptomatic peripheral vascular disease.
* Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
* Patients receiving any concomitant systemic therapy for renal cell cancer are excluded, but patients taking bisphosphonates and megestrol acetate are not excluded.
* Patients must not require total parenteral nutrition with lipids.
* Patients must not have significant proteinuria at baseline. Patients who are unexpectedly discovered to have greater than or equal to 1+ proteinuria on routine urinalysis at baseline should undergo a 24 hour urine collection, which must be an adequate collection and must demonstrate less than or equal to 1g of protein/24 hour to allow participation in the study.
* Patients must not have clinical history of coagulopathy, bleeding diathesis or thrombosis.
* Patients must not have a serious, nonhealing wound, ulcer, or bone fracture.
* Pregnancy (positive pregnancy test) or lactation.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment.
* Know hypersensitivity to any component of bevacizumab.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 22, 2005 to April 4, 2008. All participants were recruited at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the fifty-two (52), two enrolled participants did not receive treatment and were excluded from the trial.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 61 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time to progression calculated from the start of the study drug to the first evidence of disease progression. Time to progression reported as PFS measured in months. Progression (or progressive disease) defined by Response Evaluation Criteria in Solid Tumors (RECIST) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 3 years (or until disease progression)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 50
months | 11 [5.5 to 15.6]

2. Secondary Outcome: Safety of Treatment
Description: Safety measured by participant toxicities in therapy with bevacizumab for Renal Cell Carcinoma (RCC).
Time Frame: Following 56 days treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 34/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=50)
Hypertension (Blood and lymphatic system disorders) | 8
Diarrhea (Gastrointestinal disorders) | 6
Anemia (Blood and lymphatic system disorders) | 5
Fatigue (General disorders) | 6
Hyperglycemia (Blood and lymphatic system disorders) | 3
Elevated creatinine (Blood and lymphatic system disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Hypoalbuminemia (Blood and lymphatic system disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Allergic reaction (Immune system disorders) | 2
Anorexia (Gastrointestinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Thrombus/embolus (Blood and lymphatic system disorders) | 3
Wound healing delay/dehiscence (Skin and subcutaneous tissue disorders) | 2
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hemorrhage (Blood and lymphatic system disorders) | 2
Hypotension (Blood and lymphatic system disorders) | 1
Appendicitis (Infections and infestations) | 1
Neuropathy (Nervous system disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Pancreatitis (Infections and infestations) | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypokalemia (Blood and lymphatic system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Supraventricular arrhythmia (Cardiac disorders) | 1
Hyperuricemia (Blood and lymphatic system disorders) | 3
Dysarthria (Musculoskeletal and connective tissue disorders) | 1
Weight gain (General disorders) | 1
Death not associated with study drug (General disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=50)
Hypertension (Blood and lymphatic system disorders) | 38
Diarrhea (Gastrointestinal disorders) | 33
Anemia (Blood and lymphatic system disorders) | 50
Fatigue (General disorders) | 50
Hyperglycemia (Blood and lymphatic system disorders) | 50
Elevated creatinine (Blood and lymphatic system disorders) | 30
Abdominal pain (Gastrointestinal disorders) | 16
Hypoalbuminemia (Blood and lymphatic system disorders) | 21
Nausea (Gastrointestinal disorders) | 34
Bone pain (Musculoskeletal and connective tissue disorders) | 28
Vomiting (Gastrointestinal disorders) | 22
Anorexia (Gastrointestinal disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 48
Wound healing delay/dehiscence (Skin and subcutaneous tissue disorders) | 10
Hyperbilirubinemia (Blood and lymphatic system disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Hemorrhage (Blood and lymphatic system disorders) | 21
Neuropathy (Nervous system disorders) | 3
Proteinuria (Blood and lymphatic system disorders) | 33
Hyperuricemia (Blood and lymphatic system disorders) | 19
Dysarthria (Musculoskeletal and connective tissue disorders) | 6
Weight gain (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No